CLINICAL TRIAL: NCT02158494
Title: Cranial Nerve Noninvasive Neuromodulation Using the PoNS for Treatment of Symptoms Due to Mild or Moderate Traumatic Brain Injury
Brief Title: Noninvasive Neuromodulation for Treatment of Symptoms Due to Mild or Moderate Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-0002
Record Dates: First submitted 2014-05-14; First posted 2014-06-06 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Brain Injuries, Traumatic
Keywords: Cranial Nerve Noninvasive Neuromodulation; Portable Neuromodulation Stimulator (PoNS); Balance and Gait Training; Breathing Awareness Training
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurostimulation (Experimental): Balance and gait training using neurostimulation modulation. 2-week in lab training (ITP), (2 in-lab training sessions and 1 home training session daily) followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training).
  Interventions: Device: Balance and Gait Training using neurostimulation modulation.
- Minimally perceivable stimulation (Sham Comparator): Balance and gait training using non-zero, minimally perceivable stimulation (sham device). 2-week in lab training (ITP), (2 in-lab training sessions and 1 home training session daily) followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training).
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Balance and Gait Training using neurostimulation modulation. — CN-NINM uses sequenced patterns of electrical stimulation on the tongue. Our hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
  Other Names: Cranial Nerve Non-invasive Neuromodulation (CN-NINM); Portable Neuromodulation Stimulator (PoNS)
  Arms: Neurostimulation
Device: Sham Device — The sham device is visually identical to the CN-NINM device, and offers a non-zero, minimally perceivable stimulation.
  Arms: Minimally perceivable stimulation

SUMMARY:
The investigators hypothesis is that electrical stimulation to the tongue that directly stimulates two cranial nerve nuclei (Trigeminal and Facial Nerve Nuclei), will excite neural impulses to the brainstem and cerebellum. The investigators call this cranial nerve non-invasive neuromodulation (CN-NINM). The activation of these structures induces neuroplasticity when combined with specific physical, cognitive and/or mental exercises, promoting recovery of selected functional damage such as problems with balance or walking.

44 subjects will be recruited for 2 weeks of intensive In-Lab Balance and Gait Training followed by 12 weeks of intensive Home Training with weekly In-Lab check sessions. Half of the subjects will use CN-NINM in conjunction with the exercise. Half of the subjects will use very low level stimulation in conjunction with the exercise, and will serve as a control group.

DETAILED DESCRIPTION:
* Based on the results of the investigators pilot study in moderate traumatic brain injury (M-TBI), the investigators will conduct a randomized, controlled study of cranial nerve non-invasive neuromodulation (CN-NINM) in individuals with chronic symptoms of mild to moderate traumatic brain injury (mTBI), post-concussive sequelae, (PCS) and post-traumatic stress (PTS).
* The study will involve training of both balance and gait, with assessments using standardized and relevant metrics to monitor changes in these indications, as well as cognitive function, sleep, headache, anxiety, mood, and eye-movement control.
* The training regimen involves using a neurostimulation intervention that addresses primary and secondary symptoms associated with mTBI, PCS, and PTS.
* This randomized double blind controlled study will enroll a total of 44 subjects (M & F) in 2 equal subgroups: 22 with an Active PoNS™, and 22 with a Control (non-zero, minimally perceivable stimulation) device.
* Subjects will participate in a 3-phase intervention beginning with a 2-week in-lab training program (ITP) (2 in-lab training sessions and 1 home training session daily), followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training). Subjects will return to the clinic weekly during the at-home phase for a single session of retraining and progression, and participate in periodic retesting.
* All training and testing will be performed uniformly across all subjects in both groups. Multiple assessment metrics will capture data at the beginning and end of the 2-week in-lab CN-NINM intervention period and at 3-week intervals. After completion of the formal training period, subjects will stop using the device (withdrawal stage) and will be tested every 3 weeks over an additional 12 weeks to monitor and assess changes due to withdrawal of the PoNS. This will yield a total of 10 data points for each subject.
* If successful, this study would indicate that CN-NINM may improve rehabilitation outcomes and reduce time required to improve function.

ELIGIBILITY:
Inclusion Criteria:

* All candidates will have a balance disorder as a result of a traumatic brain injury (TBI).
* All candidates will have a NeuroCom® Sensory Organization Test (SOT) composite score at least 8 points below normal after adjustment for age and height [based on normative data].
* All candidates will be between the ages of 18 and 65 (at the time of screening).
* If female of childbearing potential, the candidate agrees to use adequate contraception throughout participation in the study (from enrollment to completion).
* All candidates must have access to a treadmill.
* All candidates will be at least 1 year post-injury.
* All candidates will have a neuroradiologic scan and report after their most recent TBI.
* All candidates will be ambulatory and able to walk for 20 minutes.
* All candidates, if on medications, will not have had any major changes in type or dosage within 3 months of enrollment.
* All candidates will have participated in a focused physical rehabilitation program for their TBI and feel that they have reached a plateau.
* All candidates will be able to understand and willing to give informed consent.

Exclusion Criteria:

* All candidates that have oral health problems (e.g. gum disease, active cankers, piercings, oral surgery within the previous 3 months).
* All candidates with non-removable metal orthodontic devices (e.g., braces) or oral cavity piercings that could interfere with PoNS™ use.
* All candidates who have chronic infectious diseases (e.g. hepatitis, HIV, TB).
* All candidates with unmanaged hypertension.
* All candidates with unmanaged diabetes, or complications due to diabetes (e.g. retinopathy, neuropathy, renal disease).
* All candidates with neurological disorders other than those attributed to their primary diagnosis (e.g., MS, PD, ALS, AD or other dementia, uncontrolled pain).
* All candidates with a history of oral cancer.
* All candidates who have been treated for any type of cancer other than basal cell carcinoma within the past year.
* All candidates who have had a penetrating injury, craniotomy (with the exception of a burr hole [trephination] for resolution of acute subdural hematoma), or refractory subdural hematoma.
* Exceptions for other abnormalities identified in neuroradiologic scan reports that are asymptomatic and not expected to change may be made on a case by case basis by the Medical Advisor.
* All candidates with chronic use of psychoactive or psychostimulant medications that, in the opinion of the investigators, would compromise the subject's ability to comprehend and perform the study activities.
* All candidates who have a pacemaker, or are identified as at-risk for cardiovascular events.
* All candidates who are pregnant or lactating.
* All candidates with a lower extremity biomechanical prosthetic.
* All candidates with a history of seizures (except those in the acute or post-acute phases, and are controlled).
* All candidates who who experienced a loss of consciousness greater than 24 hours as a result of their TBI.
* All candidates with a "severe" score in any of the Attention, Memory, or Executive Functions categories on the Cognitive Linguistic Quick Test (CLQT).
* All candidates who, in the opinion of the investigators, are unable to feel the stimulation and successfully complete the device level setting procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E Tyler, MS, Principal Investigator — TCNL, Department of Kinesiology, University of Wisconsin, Madison
Locations (1):
- TCNL, Department of Kinesiology, UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification will be available to researchers for independent verification of study outcomes or to conduct subsequent clinical research, whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months after publication of primary outcomes, and ending 5 years after that date.
Access Criteria: Proposals should be directed to metyler1@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- See also: related info — https://directory.engr.wisc.edu/bme/Faculty/Tyler_Mitchell/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 subjects provided consent but did not enroll in the study at sites under UW-Madison purview.
Groups:
- Control (Non-zero, Minimally Perceivable Stimulation): Balance and gait training using non-zero, minimally perceivable stimulation. 2-week in lab training (ITP), (2 in-lab training sessions and 1 home training session daily) followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training).
Period: Overall Study
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation) | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.05 (5.91) | 53.24 (10.55) | 53.89 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 19 | 20 | 39
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: NeuroCom Computerized Dynamic Posturography Sensory Organization Test (SOT)
Description: SOT assesses the ability to use visual, proprioceptive, and vestibular cues to maintain postural stability. Subjects stand on dual-force plates and the anterior-posterior sway is recorded. 6 conditions are tested (3, 20-sec trials each): Eyes open on firm surface; Eyes closed on firm surface; Eyes open with sway referenced visual surround; Eyes open on sway referenced support surface; Eyes closed on sway referenced support surface; Eyes open on sway referenced support surface and surround.
  A composite score is generated by the NeuroCom BalanceMaster System using an algorithm to calculate the composite score from each of the 3 serial repetitions for each of the 6 conditions (a total of 18 sub-scores). The calculated composite score ranges from 0 to 100 points; 0 is complete failure, 100 is perfect stability, 70 is the lower limit normal. Group mean score for each time-point is reported.
Time Frame: Baseline, 2, 14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurostimulation; Control (Non-zero, Minimally Perceivable Stimulation): This randomized double blind controlled study will enroll a total of 44 subjects (M & F) in 2 equal subgroups: 22 with an Active PoNS™, and 22 with a Control (non-zero, minimally perceivable stimulation) device. Subjects will participate in a 3-phase intervention beginning with a 2-week in-lab training program (ITP) (2 in-lab training sessions and 1 home training session daily), followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training). Subjects will return to the clinic weekly during the at-home phase for a single session of retraining and progression, and participate in periodic retesting.
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
score on a scale
  Baseline | 42.77 (17.54) | 36.24 (16.09)
  Week 2 | 63.73 (15.06) | 62.00 (22.32)
  Week 14 | 70.89 (11.45) | 71.21 (16.95)
  Week 26 | 74.83 (11.86) | 71.50 (17.50)
Statistical Analysis 1: Comparison: Neurostimulation vs Control (Non-zero, Minimally Perceivable Stimulation); P-Value for Sensory Organization Test results at 2 weeks; Test type: Superiority; p = 0.41, t-test, 2 sided
Statistical Analysis 2: Comparison: Neurostimulation vs Control (Non-zero, Minimally Perceivable Stimulation); P-Value for Sensory Organization Test results at 14 weeks; Test type: Superiority; p = 0.47, t-test, 2 sided
Statistical Analysis 3: Comparison: Neurostimulation vs Control (Non-zero, Minimally Perceivable Stimulation); P-Value for Sensory Organization Test results at 26 weeks; Test type: Superiority; p = 0.99, t-test, 2 sided

2. Other Pre Specified Outcome: Change in Neurobehavioral Symptom Inventory Over Baseline
Description: A 22-item subjective inventory of TBI symptoms where symptoms are scored on a scale of 0 (none) to 4 (very severe). Lower scores indicate decreased symptoms. Group mean change from baseline at 2, 14, and 26 weeks is reported. The range of possible scores if from 0 to 88. The results are reported as a change from baseline.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
score on a scale
  Week 2 | -13.52 (9.17) | -7.52 (13.58)
  Week 14 | -10.47 (10.12) | -7.10 (9.83)
  Week 26 | -9.94 (15.49) | -8.40 (10.46)

3. Other Pre Specified Outcome: Change in 6-Minute Walk Test (6MWT) Over Baseline
Description: Measures walking speed over ground. The six-minute walk test (6MWT) measures the distance in meters an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. Change in 6MWT over baseline for each time point is reported.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
meters
  Week 2 | 33.06 (75.01) | 19.02 (39.41)
  Week 14 | 72.27 (79.97) | 62.30 (51.04)
  Week 26 | 76.81 (95.41) | 74.38 (49.21)

4. Other Pre Specified Outcome: Change in Dynamic Gait Index (DGI) Over Baseline
Description: Assesses walking, walking with head turns, over and around obstacles, and stairs. Dynamic Gait Index - A semiquantitative tool used to evaluate a patient's ability to modify gait by changing task demands, esp. in patients with dizziness and balance deficits. This test is used to identify patients, esp. older adults, who are predisposed to falling. Participants are graded from 0 (low function) to 3 (high function) on 8 tasks: normal walking, their ability to vary walking speed, turn their heads, turn their bodies, step over and around obstacles, climb stairs, turn while walking. The range of scores is 0-24, higher scores indicate higher function, with a score of 24 considered Normal. Change from baseline to 2, 14, and 26 weeks is reported.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurostimulation: Balance and gait training using neurostimulation modulation. 2-week in lab training (ITP), (2 in-lab training sessions and 1 home training session daily) followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training).
  Balance and Gait Training using neurostimulation modulation.: Cranial-nerve Non-invasive Neuromodulation (CN-NINM) uses sequenced patterns of electrical stimulation on the tongue. Our hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
- Minimally Perceivable Stimulation: Balance and gait training using non-zero, minimally perceivable stimulation. 2-week in lab training (ITP), (2 in-lab training sessions and 1 home training session daily) followed by 12 weeks of training at home (HTP) (3 home training sessions daily), and a 12-week withdrawal period (no training).
  Balance and Gait Training using neurostimulation modulation.: CN-NINM uses sequenced patterns of electrical stimulation on the tongue. Our hypothesis is that CN-NINM induces neuroplasticity by noninvasive stimulation of two major cranial nerves: trigeminal, CN-V, and facial, CN-VII.
Arm/Group | Neurostimulation | Minimally Perceivable Stimulation
Number analyzed (Participants) | 22 | 21
score on a scale
  Week 2 | 2.23 (2.88) | 1.76 (2.72)
  Week 14 | 3.58 (3.53) | 3.42 (3.11)
  Week 26 | 4.12 (3.67) | 3.45 (3.41)

5. Other Pre Specified Outcome: Change in California Verbal Learning Test (CVLT) Over Baseline
Description: Assesses short- and long-term verbal memory by evaluating a series of recall and recognition tasks. The test is scored via computer algorithm. A score of 50 represents is equal to the population mean, the normal range is between 40-60 (ie. +/- 1 SD from the mean). The total range of possible scores is 0 (no recalled words) to 100 (all correct). Change in score over baseline at 2, 14, and 26 weeks is reported.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
units on a scale
  Week 2 | 8.95 (8.48) | 9.71 (6.63)
  Week 14 | 9.00 (11.34) | 11.30 (9.40)
  Week 26 | 10.28 (11.79) | 11.00 (9.70)

6. Other Pre Specified Outcome: Change in Brief Symptom Inventory 18 (BSI 18) Over Baseline
Description: A short, reliable, 18-question instrument for assessment of psychological distress (anxiety, depression, & somatization) in a clinical population. It is scored from 0-4, with a total range of possible scores 0-72 where higher scores indicate more distress.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurostimulation | Minimally Perceivable Stimulation
Number analyzed (Participants) | 22 | 21
units on a scale
  Week 2 | -5.32 (9.10) | -2.38 (7.53)
  Week 14 | -4.16 (9.41) | -2.95 (6.13)
  Week 26 | -7.72 (10.15) | -2.50 (6.93)

7. Other Pre Specified Outcome: Change in Wechsler Adult Intelligence Scale - Symbol Search and Coding (WAIS-IV) Over Baseline
Description: Assesses visual spatial abilities. The Symbol Search and Coding WAIS-IV subtests measure Processing Speed, an indicator of the rate of cognitive processing and creating an appropriate response output. The tasks require attending to visual material, visual scanning and perception, spatial organization, hand-eye coordination, and paired associative learning. The raw score (processing speed for each test) is converted to a scaled score 1-10 for each and summed for a total possible score of 2-20, the higher the score, the more improved the processing speed. Change in score from baseline to 2, 14, and 26 weeks are reported.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
score on a scale
  Week 2 | 0.95 (2.38) | 1.14 (2.29)
  Week 14 | 1.11 (2.90) | 1.25 (2.02)
  Week 26 | 1.78 (2.44) | 1.20 (2.35)

8. Other Pre Specified Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline
Description: Subjective inventory of sleep habits, duration and quality. It is scored from 7 components (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction) to provide a global PSQI score. Most items are scored from 0-3 where 3 is a negative extreme, therefore lower cumulative scores are indicative of improved sleep habits. The total range of scores is from 0-21.
Time Frame: Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
score on a scale
  Baseline | 9.318 (4.874) | 9.182 (4.934)
  Week 2 | 8.682 (5.213) | 7.810 (5.698)
  Week 14 | 8.611 (4.742) | 8.714 (5.349)
  Week 26 | 8.294 (5.084) | 8.238 (5.272)

9. Other Pre Specified Outcome: Change in Headache Disability Index (HDI) From Baseline
Description: Assesses frequency & severity of headaches via a 25-item questionnaire where an answer of 'yes' = 4 points, 'sometimes' = 2 points, and 'no' = 0 points. The lower the score, the less frequent and severe the symptoms. The range of possible scores is 0 to 100. The results are reported as a change from baseline.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurostimulation | Control (Non-zero, Minimally Perceivable Stimulation)
Number analyzed (Participants) | 22 | 21
score on a scale
  Week 2 | -16.00 (23.56) | -4.38 (20.15)
  Week 14 | -9.79 (18.02) | -11.00 (20.62)
  Week 26 | -14.78 (21.17) | -13.60 (23.48)

10. Other Pre Specified Outcome: Electromyography (EMG)
Description: Measures muscle activation patterns during gait.
Time Frame: Change from Baseline at 2,14, and 26 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Computerized Video Nystagmography (VNG)
Description: Measures eye movement control under 3 static (x and y axis fixation, spontaneous nystagmus), and 3 dynamic conditions (random saccade, smooth pursuit, optokinetic nystagmus).
Time Frame: Change from Baseline at 2,14, and 26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: * Category - the medical terminology for the adverse event or unanticipated problem category from the Safety Profiler list of Common Terminology Criteria for Adverse Events (http://safetyprofiler-ctep.nci.nih.gov/CTC/CTC.aspx)
  * AE Detail - a detailed description of the severity of the category from the Safety Profiler list of Common Terminology Criteria for Adverse Events (http://safetyprofiler-ctep.nci.nih.gov/CTC/CTC.aspx)
Arm/Group | Neurostimulation | Minimally Perceivable Stimulation
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/22 | 1/21
Other Adverse Events (participants affected / at risk) | 11/22 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurostimulation (N=22) | Minimally Perceivable Stimulation (N=21)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Subject became nauseous, with a high fever and impaired balance.Responders brought her to the hospital. She was admitted, assessed and treated. No definite cause for her symptoms was identified. All symptoms have resolved and there was no recurrence.
Gallbladder Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) — Subject was admitted to the hospital with abdominal pain and had an ultrasound of his gall bladder that showed gall stones in the gall bladder. He had surgery to remove his gall bladder. He was discharged and was given oxycodone for pain management.
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) — Subject reported that he had kidney stones. He was in the hospital for 6 days due to the kidney stones. He went into septic shock. He was treated with IV antibiotics and a stent was placed. Extracorporeal shock wave lithotripsy was scheduled.
Prostate cancer (Renal and urinary disorders) | 0 (0) | 1 (1) — During end of study wrap up, subject reported that he had been diagnosed with prostate cancer on 11 Feb 2016. He is under the care of an oncologist and was scheduled for surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurostimulation (N=22) | Minimally Perceivable Stimulation (N=21)
General Pain (General disorders) | 1 (1) | 1 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (6)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 0 (0) | 1 (2)
Diabetic Shock (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting and Diahrrea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02158494/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02158494/SAP_001.pdf